CLINICAL TRIAL: NCT00659984
Title: A Phase 2a Study of Ultratrace™ Iobenguane I 131 in Patients With Relapsed/Refractory High-Risk Neuroblastoma
Brief Title: N2007-01: Ultratrace™ Iobenguane I 131 in Patients With Relapsed/Refractory High-Risk Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593357; NANT-2007-01 (Other: NANT Consortium)
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Intervention Model Description: Ultratrace™ Iobenguane I 131
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultratrace™ Iobenguane I 131 (Experimental): Eligible patients received a diagnostic imaging dose of Ultratrace™ Iobenguane I 131 (1-5 mCi) within 7 days of study enrollment, followed by three dosimetry scans over 3-6 days. If the imaging dose demonstrated normal biodistribution and tumor uptake, then the patient received a therapeutic dose within 7-28 days of the diagnostic imaging dose, followed by a single imaging scan on Day 7 post therapy. As per protocol, therapeutic dosing was to begin at 12.0 mCi/kg and escalate to 15.0, 18.0, and 21.0 mCi/kg until the MTD was established or the 21.0 mCi/kg dose level was reached. Actual doses administered ranged from 8.8 to 18.6 mCi/kg. Based on actual doses administered, patients were grouped into 3 mean dose groups: 11.2, 15.5, and 18.2 mCi/kg.
  The dosimetry dose was administered over a period of 1-3 minutes by injection; the therapeutic dose was diluted in up to 25 mL normal saline and infused intravenously over 30 to 60 minutes.
  Interventions: Drug: UltratraceTM Iobenguane I 131 Imaging; Drug: UltratraceTM Iobenguane I 131 Therapy

INTERVENTIONS:
Drug: UltratraceTM Iobenguane I 131 Imaging — 0.1 mCi/kg [3.7 MBq/kg] (minimum dose 1mCi [37MBq] but not to exceed 5 mCi [185 MBq]) of UltratraceTM Iobenguane I 131 given 7 -28 days before therapeutic dose administration on day 0. Thyroid protection will be administered per institutional protocol for I-131-MIBG however, thyroid blocking must be started prior to the Ultratrace imaging dose. Anterior and posterior whole body images will be taken to assess organ distribution, tumor uptake and dosimetry calculations.
  Other Names: Azedra
Drug: UltratraceTM Iobenguane I 131 Therapy — Therapeutic dose will be given on Day 0 if dosimetry scans showed that the prescribed or adjusted dose will not exceed > 23 Gy to the kidneys, > 30 Gy to the liver, or > 15 Gy to the lungs. and tumor uptake confirmed with UltratraceTM imaging dose. Only one treatment course of therapeutic UltratraceTM will be given in this study.
  Other Names: Azedra

SUMMARY:
RATIONALE: Radioactive drugs, such as iodine I 131 metaiodobenzylguanidine (MIBG), may carry radiation directly to tumor cells and not harm normal cells. A bone marrow or peripheral stem cell transplant using stem cells from the patient may be able to replace blood-forming cells that were destroyed by I 131 MIBG.

PURPOSE: This phase II trial is studying the side effects and best dose of iodine I 131 MIBG followed by a stem cell transplant in treating young patients with relapsed or refractory high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum tolerated dose of iodine I 131 metaiodobenzylguanidine (^131I-MIBG) in patients with relapsed/refractory high-risk neuroblastoma.

Secondary

* To describe toxicity following treatment with ^131I-MIBG in patients with relapsed/refractory high-risk neuroblastoma.
* To estimate radiation absorbed doses to measurable lesions and to a standard set of normal organs following a 0.1 mCi/kg [3.7 MBq/kg] (minimum dose of 1.0 mCi [37 MBq] but not to exceed 5.0 mCi [185 MBq]) intravenous administration of ^131I-MIBG in patients with relapsed/refractory high-risk neuroblastoma.
* To describe, within the confines of a phase IIa trial, objective tumor response following treatment with ^131I-MIBG in patients with relapsed/refractory high-risk neuroblastoma.
* To explore dose-response following treatment with ^131I-MIBG in patients with relapsed/refractory high-risk neuroblastoma.
* To explore quality of life assessment following treatment with ^131I-MIBG in patients with relapsed/refractory high-risk neuroblastoma.

OUTLINE:

* Dosimetry: Patients receive a dosimetric dose of iodine I 131 metaiodobenzylguanidine (^131I-MIBG) IV over 1-3 minutes. Patients then undergo 2 or 3 MIBG scans within 5 days of the dosimetry dose to assess biodistribution and tumor uptake. Patients with normal tumor uptake and biodistribution proceed to treatment.
* Treatment: Within 1-4 weeks of the dosimetric dose, patients with normal tumor uptake and biodistribution receive a therapeutic dose of ^131I-MIBG IV over 1 hour on day 0 and undergo MIBG scan on day 7. Patients then proceed to autologous stem cell infusion.
* Autologous stem cell infusion: Patients receive an infusion of autologous stem cells from peripheral blood or bone marrow on day 14. Patients with an ANC of < 500/µl at any point after autologous stem cell infusion receive filgrastim (G-CSF) IV or subcutaneously once daily until ANC is > 2,000/µl.

Patients complete a quality of life questionnaire at baseline and then at day 60.

After completion of study treatment, patients are followed at day 60 and periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least one year and no more than 30 years of age when registered on this study.
* Patients must have high risk neuroblastoma and either have tumor left after treatment started at diagnosis or have had the tumor grow back (relapsed) after getting some treatment
* Patients must an MIBG scan done and it must be positive for neuroblastoma.
* Patients must have a PBSC or bone marrow stem cell product available that meets study criteria. If they don't already have stem cells frozen away then they must be able to have a stem cell pheresis done to collect the necessary amount of stem cells for study entry and these stem cells must meet study criteria.
* Patients must have adequate heart, lung, liver, kidney and bone marrow function.

Exclusion Criteria:

* They have had a stem cell transplant using another person as the stem cell donor. (You can still be in the study if a previous transplant used your own stem cells)
* They have other medical problems that could get much worse if they had this treatment.
* They are on dialysis for badly working kidneys or have other kidney problems.
* They are pregnant or breast feeding.
* They have tumor in the brain or spinal cord that is seen on a CT or MRI scan one month before starting treatment
* They had total body radiation or radiation to the entire belly.
* They have a known allergy to MIBG, iodine or SSKI.
* They can't cooperate with the special precautions that are needed during UltratraceTM MIBG treatment or with other safety monitoring requirements of the study..

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine K. Matthay, MD, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (8):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultratrace™ Iobenguane I 131: Eligible patients received a diagnostic imaging dose of Ultratrace™ Iobenguane I 131 within 7 days (d) of enrollment, followed by 3 dosimetry scans over 3-6 days. For the imaging dose, 0.1 mCi/kg (3.7 MBq/kg), at a min dose of 1 mCi (37 MBq) but not to exceed 5 mCi (185 MBq) of Ultratrace™ Iobenguane I 131 was administered 7-28 d prior to the therapeutic dose on Day 0. If the imaging dose demonstrated NL biodistribution/tumor uptake, pts received a therapeutic dose within 7-28 d of the imaging dose followed by a single imaging scan on Day 7 post therapy.
  Therapeutic dosing was to begin at 12.0 mCi/kg and escalate to 15.0, 18.0, and 21.0 mCi/kg until the MTD was established or the 21.0 mCi/kg dose level was reached. Based on actual doses administered, pts were grouped into 3 mean dose groups: 11.2, 15.5, and 18.2 mCi/kg.
  The dosimetry dose was administered over 1-3 mins by injection; the therapeutic dose was diluted in up to 25 mL normal saline and infused over 30 to 60 mins.
Period: Overall Study
Arm/Group | Ultratrace™ Iobenguane I 131
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Ultratrace™ Iobenguane I 131: Eligible patients received a diagnostic imaging dose of Ultratrace™ Iobenguane I 131 (1-5 mCi) within 7 days of study enrollment, followed by three dosimetry scans over 3-6 days. If the imaging dose demonstrated normal biodistribution and tumor uptake, then the patient received a therapeutic dose within 7-28 days of the diagnostic imaging dose, followed by a single imaging scan on Day 7 post therapy. Therapeutic dosing began at 12.0 mCi/kg and escalated to 15.0, 18.0, and 21.0 mCi/kg until the MTD was established or the 21.0 mCi/kg dose level was reached. The dosimetry dose was administered over a period of 1-3 minutes by injection; the therapeutic dose was diluted in up to 25 mL normal saline and infused intravenously over 30 to 60 minutes.
Arm/Group | Ultratrace™ Iobenguane I 131
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 8 [3 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The maximum tolerated dose (MTD) was defined as the dose immediately below the level at which dose escalation would be stopped due to dose limiting toxicities (DLTs). Once the MTD was reached, an additional 3 patients were to be treated at that dose level, for a total of 6 patients at that planned dose level. DLTs were defined as any of the events that are possibly, probably or definitely attributable to UltratraceTM iobenguane I 131. The MTD was supposed to be the highest dose tested at which fewer than 1/3 of pts experience a DLT when 6 patients have been treated at the MTD but the dosimetry results indicated that the maximal dosage allowed to normal organs would be exceeded if the highest planned dose (21.0 mCi/kg) was administered, so the highest dose administered in the study was 18.6 mCi/kg .
Time Frame: Day 60 +/-10 or Engraftment, whichever comes first
Population: A total of 15 patients underwent dosimetry (received a single imaging dose of Ultratrace™ Iobenguane I 131 injection) and all 15 patients later received a single therapeutic dose of Ultratrace™ Iobenguane I 131.
Measure: Number; unit: mCi/kg
Groups:
- Ultratrace™ Iobenguane I 131: Following therapeutic dosing at the 12.0, 15.0, and 18.0 mCi/kg cohorts, 4 patients who were to receive the 21.0 mCi/kg therapeutic dose were required to have their planned dose reduced below the dose that was calculated based on the patient's dosimetry results, in order to meet the protocol guidelines for maximal dosage allowed to normal organs described above. Because of the differences between the planned and actual therapeutic doses that were administered to several patients, patients were grouped and the study data were presented and analyzed by actual doses rather than by the planned dose cohorts of 12.0, 15.0, 18.0, and 21.0 mCi/kg. Based on the actual doses administered, patients were grouped into 3 dose groups of 6, 3, and 6 patients, according to the mean doses of the groups, which were 11.2, 15.5, and 18.2 mCi/kg, respectively.
Arm/Group | Ultratrace™ Iobenguane I 131
Number analyzed (Participants) | 15
mCi/kg | 18.6

2. Secondary Outcome: Dose Limiting Toxicities
Description: Dose limiting toxicities include treatment emergent adverse events (TEAEs) that were possibly, probably, or definitely related to Ultratrace™ Iobenguane I 131.
Time Frame: From the time of signed informed consent until Day 60 or until the end of therapy evaluation is completed (whichever comes first).
Population: as for outcome 1
Measure: Number; unit: number of DLTs
Groups:
- 11.2 mCi Group: 11.2 mCi/kg Ultratrace™ Iobenguane I 131 represents the mean dose administered to this group of subjects.
- 15.5 mCi Group: 15.5 mCi/kg Ultratrace™ Iobenguane I 131 represents the mean dose administered to this group of subjects.
- 18.2 mCi Group: 18.2 mCi/kg Ultratrace™ Iobenguane I 131 represents the mean dose administered to this group of subjects.
Arm/Group | 11.2 mCi Group | 15.5 mCi Group | 18.2 mCi Group
Number analyzed (Participants) | 6 | 3 | 6
number of DLTs | 0 | 0 | 0

3. Secondary Outcome: Dosimetric Estimation of Radiation Absorbed Doses to Measurable Lesions
Description: The dosimetric endpoint was to estimate radiation absorbed doses to measurable lesions and to a standard set of normal organs following an imaging dose of 0.1 mCi/kg Ultratrace™ Iobenguane I 131. Biodistribution was assessed by determination of total body residence (TBR) time and by visual examination of whole body camera images. 3 timepoints were used, the 1st image was taken within 1hr after the imaging dose, the 2nd image was taken at ~24hr after imaging dose, the 3rd image was taken 2-5d after imaging dose. Whole body radiation absorbed dose estimates & kidney, liver, and lung were calculated using the Medical Internal Radiation Dose (MIRD) schema.TBR time is derived from time integration of curve-fitted injected activity across all 3 timepoints when the isotope is emitting radiation.Three points are sampled to estimate a singular value for each organ and tissue according to the commonly used methods of the Society of Nuclear Medicine and Molecular Imaging Committee on MIRD.
Time Frame: Day 5 post Dosimetric Dose
Population: A total of 15 patients underwent dosimetry (received a single imaging dose of Ultratrace™ Iobenguane I 131 injection).
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Ultratrace™ Iobenguane I 131
Number analyzed (Participants) | 15
Gy
  Kidney | 16.7 (5.2)
  Liver | 12.7 (4.1)
  Lungs | 11.1 (2.8)

4. Secondary Outcome: Overall Objective Tumor Response Post Therapeutic Treatment
Description: The International Neuroblastoma Response Criteria (INRC) were utilized as a basis for the overall response criteria, which incorporated responses in MIBG positive lesions,bone marrow disease, and CT/MRI lesions that met NANT-modified RECIST criteria. Efficacy success was defined as the proportion of pts who were successful overall [i.e., achieving a Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR)] determined by independent reviewers. CR = Disappearance of all target lesions, homovanillic acid/ vanillylmandelic acid (HVA/VMA) normal (NL); VGPR = > 90% decr of disease for CT/MRI target lesions, all pre-existing bone lesions with CR by MIBG; MIBG scan can be SD/CR in soft tissue lesions. CR in bone marrow, no new tumor sites, and NL HVA/VMA.; PR = At least 30% decr in disease measurement for CT/MRI target lesions. Bone marrow with CR, MIBG with either PR/CR in bone lesions, MIBG may be SD /CR in soft tissue lesions, and HVA/VMA may still be elevated.
Time Frame: Day 60 +/- 10 days post Therapeutic Dose
Population: The evaluable population (which excludes non-evaluable responses) contains one patient less than the full ITT population.
Measure: Number (95% Confidence Interval); unit: proportion of evaluable population
Groups:
- Ultratrace™ Iobenguane I 131: The proportion of patients who were considered successful defined as a patient achieving a Complete Response, Very Good Partial Response or Partial Response as determined by the Independent Reviewers.
Arm/Group | Ultratrace™ Iobenguane I 131
Number analyzed (Participants) | 14
proportion of evaluable population | 0.29 [0.01 to 0.56]

5. Secondary Outcome: Tumor Response in CT/MRI Lesions Post Therapeutic Treatment
Description: Measurable disease was defined for a conventional CT scan by the presence of at least one lesion that could be accurately measured in at least one dimension with the longest diameter at least 20 mm by Independent Review. Efficacy success was defined as a patient achieving a Complete Response (CR)=disappearance of all target and non-target CT/MRI lesions; or, Very Good Partial Response (VGPR)=greater than 90% decrease of the disease measurement for CT/MRI lesions, taking as reference the disease measurement done to confirm measurement disease at study entry. Non-target CT/MRI lesions stable to smaller in size; or, Partial Response (PR)=at least 30% decrease in the disease measurement for CT/MRI lesions, taking as reference the disease measurement done to confirm measurable disease at study entry. Non-target CT/MRI lesions stable to smaller in size.
Time Frame: Day 60 +/- 10 days post Therapeutic Dose
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of evaluable population
Groups:
- Over Tumor Response: The proportion of patients who were considered successful defined as a patient achieving a Complete Response, Very Good Partial Response or Partial Response as determined by the Independent Reviewers.
Arm/Group | Over Tumor Response
Number analyzed (Participants) | 14
percentage of evaluable population | 21 [0 to 46]

6. Secondary Outcome: Quality of Life
Description: Patients (aged 5-18) and parents (of patients aged 2-18) were asked to complete the 23-item Pediatric Quality of Life InventoryTM (PedsQLTM). PedsQLTM consists of 4 scales (physical, emotional, social, school functioning) which are then averaged into an overall summary score (scale: 0-100 with 0 representing the worst possible Quality of Life overall summary score and 100 representing the best possible Quality of Life overall summary score). The mean difference between the post treatment overall summary score and the baseline overall summary score is reported.
Time Frame: Day 60 +/- 10 days post Therapeutic Dose
Population: Self reported PedsQL™ scores were obtained for 9 patients in the ITT population (n=15) at baseline (prior to the start of the Ultratrace™ Iobenguane I 131 imaging studies) and at the end of therapy (60 ±10 days post treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ultratrace™ Iobenguane I 131: Based on the actual doses administered, patients were grouped into 3 dose groups of 6, 3, and 6 patients, according to the mean doses of the groups, which were 11.2, 15.5, and 18.2 mCi/kg, respectively.
Arm/Group | Ultratrace™ Iobenguane I 131
Number analyzed (Participants) | 9
units on a scale | 5.2 (11.27)
Statistical Analysis 1: Comparison: Ultratrace™ Iobenguane I 131; Test type: Superiority or Other; p = 0.363, Cochran Armitage Trend Test; Hazard Ratio (HR) = 5.2, 95% CI 2-sided [-3.4 to 13.9]

ADVERSE EVENTS:
Time Frame: From the time of signed informed consent until Day or until the end of therapy evaluation was completed (whichever occurred first).
Description: Serious adverse events (SAEs) that were ongoing at study completion (Day 60 ±10 days) were followed for 60 days or until resolution, whichever occurred first.
Groups:
- Ultratrace™ Iobenguane I 131: Eligible patients received a diagnostic imaging dose of Ultratrace™ Iobenguane I 131 (1-5 mCi) within 7 days of study enrollment, followed by three dosimetry scans over 3-6 days. If the imaging dose demonstrated normal biodistribution and tumor uptake, then the patient received a therapeutic dose within 7-28 days of the diagnostic imaging dose, followed by a single imaging scan on Day 7 post therapy. Mean therapeutic dosing groups were 11.2 mCi/kg, 15.5 nCi/kg and 18.2 mCi/kg. The dosimetry dose was administered over a period of 1-3 minutes by injection; the therapeutic dose was diluted in up to 25 mL normal saline and infused intravenously over 30 to 60 minutes.
Arm/Group | Ultratrace™ Iobenguane I 131
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultratrace™ Iobenguane I 131 (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Disease progression (General disorders) | 1 (1)
Neutropenia infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultratrace™ Iobenguane I 131 (N=15)
Leukopenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 8
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Aspartate aminotransferase increased (Investigations) | 12
Hemoglobin decreased (Investigations) | 11
Alanine aminotransferase increased (Investigations) | 9
Activated partial thromboplastin time prolonged (Investigations) | 3
Blood bilirubin increased (Investigations) | 3
Weight decreased (Investigations) | 3
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Salivary gland pain (Gastrointestinal disorders) | 4
Salivary gland enlargement (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Pyrexia (General disorders) | 5
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Candidiasis (Infections and infestations) | 2
Headache (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 2
Bladder spasm (Renal and urinary disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less